CLINICAL TRIAL: NCT04530526
Title: Surgical Treatment of Post-surgical Mastectomy Pain Utilizing the Regenerative Peripheral Nerve Interface (RPNI)
Brief Title: Surgical Treatment of Post-surgical Mastectomy Pain Utilizing the Regenerative Peripheral Nerve Interface
Acronym: RPNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.124; HUM00149189 (Other: University of Michigan); R21CA234760 (NIH)
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Post-Mastectomy Chronic Pain Syndrome
Keywords: neuroma,outcome-assessment health care, post-mastectomy; outcome-assessment health care; post-mastectomy; neuroma
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regenerative Peripheral Nerve Interface (RPNI) (Other): Using evaluative ultrasound measurements and a standard panel of patient-reported outcome measures (PROMs) to measure pain experience, anxiety and depression, patients will be evaluated at baseline (T1=0months), pre-operatively following 3 months of standard neuropathic pain management therapy (T2=3months) and at three months (T3=6months) and nine months (T4=12months) post RPNI surgery.
  Interventions: Procedure: Regenerative Peripheral Nerve Interface

INTERVENTIONS:
Procedure: Regenerative Peripheral Nerve Interface — The regenerative peripheral nerve interface (RPNI) has emerged as a novel strategy to treat neuromas in peripheral nerves. The RPNI consists of the residual peripheral nerve end implanted in a skeletal muscle graft, following surgical resection of the injured terminal nerve portion (neuroma). The free muscle graft is separated from its native nerve innervation, leaving open neuromuscular junctions for ingrowth and attachment of nerve fibers from the implanted nerve.

SUMMARY:
Post-mastectomy pain due to nerve injury leads to long-term opioid use and diminished quality-of-life. The investigators on this study will evaluate the regenerative peripheral nerve interface (RPNI), a novel surgical approach to neuroma treatment, to improve patient-reported post-mastectomy pain and definitively treat intercostal neuromas after mastectomy.

DETAILED DESCRIPTION:
Up to 40% of patients who undergo mastectomy suffer from chronic pain, defined as pain lasting greater than three months. Chronic post-mastectomy pain due to nerve injury leads to long-term opioid use and diminished quality-of-life. A novel surgical approach to neuroma treatment, the regenerative peripheral nerve interface (RPNI) developed to treat painful neuromas associated with limb amputation has shown significant reductions in patient-reported pain. RPNI surgery is now available through Michigan Medicine's Multi-Disciplinary Peripheral Nerve (MDPN) Clinic to improve post-mastectomy pain and definitively treat intercostal neuromas following mastectomy. Using patient-reported outcomes and clinical data the investigators will evaluate the use of RPNI surgery to reduce persistent post- mastectomy pain in women seeking surgical consultation through the Plastic Surgery or MDPN clinics.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Reporting post-mastectomy pain at least six months removed from mastectomy or partial mastectomy (lumpectomy).
* Willing to comply with all study procedures and be available for the duration of the study
* Fluent in English
* Women of reproductive potential must use highly effective contraception (specify methods of contraception acceptable for the study, e.g., licensed hormonal methods) and/or willingness to undergo a pregnancy test.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Previous surgical management for chronic post-mastectomy pain
* Signs/symptoms which are not suggestive of neuropathic pain based on physical exam at time of consultation.
* Pregnancy or lactation
* Men will not be enrolled in this study due to the low prevalence of male mastectomy.
* Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Brown, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nag S, Kennedy P, Aris K, Moore AM, Farhadi R. The Role of Nerve Surgery in the Management of Post-Breast Surgery Pain Syndrome: A Systematic Review and Meta-analysis. Ann Plast Surg. 2025 Dec 1;95(6):625-629. doi: 10.1097/SAP.0000000000004516. Epub 2025 Oct 16. PMID 41133892

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Started | 26
Completed | 20
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 26
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 1
  40-49 years | 9
  50-59 years | 5
  60-69 years | 8
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level
Description: The use of RPNI surgery to reduce post-mastectomy pain will be evaluated by validated patient-reported outcome (PRO) surveys administered at 4 timepoints: at baseline (at time of enrollment), at the RPNI pre-operative visit (approximately 3 months after enrollment), and at approximately 3 and 9 months after RPNI surgery. The average time of study involvement for each patient will be 12 months. Patients enrolled during the first year of the study's 2-year recruitment period may be followed until the study stops.
  Numerical Pain Rating Scale (0-10)- 10 indicating more pain Short Form McGill Pain Questionnaire 2 (0-10)- 10 indicating more pain Pain Catastrophizing Score (0-52)- 52 indicating more pain PROMIS Intensity (0-12)- 12 indicating more pain PROMIS Interference (0-24)- 24 indicating more pain PROMIS Neuropathic (0-20)- 20 indicating more pain
Time Frame: baseline, and 9 months post surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 20
score on a scale
  Numerical Pain Rating Scale- Preoperative Score | 6.9 (0.4)
  Numerical Pain Rating Scale- Postoperative Score | 0.6 (0.3)
  Short Form McGill Pain Questionnaire 2- Preoperative | 4.4 (0.5)
  Short Form McGill Pain Questionnaire 2- Postoperative | 2.5 (0.6)
  Pain Catastrophizing Score- Preoperative | 27.5 (3.0)
  Pain Catastrophizing Score- Postoperative | 14.1 (2.9)
  PROMIS Intensity- Preoperative | 7.9 (0.5)
  PROMIS Intensity- Postoperative | 4.9 (0.8)
  PROMIS Interference- Preoperative | 16.2 (1.3)
  PROMIS Interference- Post Operative | 11.0 (2.0)
  PROMIS Neuropathic- Preoperative | 8.6 (1.4)
  PROMIS Neuropathic- Postoperative | 6.0 (1.4)

2. Primary Outcome: Change in Depression/Anxiety Scores
Description: Evaluated by validated patient-reported outcome (PRO) surveys administered at 4 timepoints: at baseline (at time of enrollment), at the RPNI pre-operative visit (approximately 3 months after enrollment), and at approximately 3 and 9 months after RPNI surgery. The average time of study involvement for each patient will be 12 months. Patients enrolled during the first year of the study's 2-year recruitment period may be followed until the study stops.
  Patient Health Questionnaire-9 range is 0-27. 27 indicates a worse outcome. Generalized Anxiety Disorder-7 range is 0-21. 21 indicates a worse outcome.
Time Frame: baseline, and 9 months post surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 20
score on a scale
  Patient Health Questionnaire-9- Preoperative | 10.3 (1.3)
  Patient Health Questionnaire-9- Postoperative | 7.2 (1.4)
  Generalized Anxiety Disorder-7- Preoperative | 7.3 (1.1)
  Generalized Anxiety Disorder-7- postoperative | 4.3 (1.2)

3. Primary Outcome: Change in Opioid Consumption (Number of Opioid Medications)
Description: Evaluated by validated patient-reported outcome (PRO) surveys administered at 4 timepoints: at baseline (at time of enrollment), at the RPNI pre-operative visit (approximately 3 months after enrollment), and at approximately 3 and 9 months after RPNI surgery. The average time of study involvement for each patient will be 12 months. Patients enrolled during the first year of the study's 2-year recruitment period may be followed until the study stops.
Time Frame: baseline, and 9 months post surgery
Measure: Mean (Standard Error); unit: Opioid medications
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 20
Opioid medications
  Number of Opioid Medications- Preoperative | 1.3 (0.2)
  Number of Opioid Medications- Postoperative | 0.4 (0.2)

4. Primary Outcome: Freedom From Neuroma Recurrence Evaluated by Physical Exam
Description: Data will be derived from standard clinical care for patients seeking surgical management of post-mastectomy chronic pain. Physical examinations will be performed at the time of patient enrollment and subsequent follow-up visits, as part of routine clinical evaluation, up to approximately 9 months after RPNI surgery. Patients enrolled during the first year of the study's 2-year recruitment period may be followed until the study stops.
Time Frame: 24 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 20
Participants | 20

5. Primary Outcome: Freedom From Neuroma Recurrence Evaluated by Ultrasound
Description: Data will be derived from standard clinical care for patients seeking surgical management of post-mastectomy chronic pain. Ultrasound will be performed at the time of patient enrollment and subsequent follow-up visits, as part of routine clinical evaluation, up to approximately 9 months after RPNI surgery. Patients enrolled during the first year of the study's 2-year recruitment period may be followed until the study stops.
Time Frame: 24 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 20
Participants | 20

6. Primary Outcome: Change in Opioid Consumption (Oral Morphine Equivalents)
Description: as for outcome 3
Time Frame: baseline, and 9 months post surgery
Measure: Mean (Standard Error); unit: mg morphine equivalent
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
Number analyzed (Participants) | 20
mg morphine equivalent
  Oral Morphine Equivalents (mg)- Preoperative | 43.3 (11.4)
  Oral Morphine Equivalents (mg)- Postoperative | 12.0 (4.9)

ADVERSE EVENTS:
Time Frame: There is minimal perceived risk associated with this study and adverse events were not collected.
Description: There is minimal perceived risk associated with this study and adverse events were not collected.
Arm/Group | Regenerative Peripheral Nerve Interface (RPNI)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04530526/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT04530526/ICF_000.pdf